CLINICAL TRIAL: NCT05532631
Title: Percutaneous Coronary RevascularizatiOn VERsus Coronary-Artery Bypass Grafting for Multivessel Disease in Patients With Left Ventricular Dysfunction (PROVERB)
Acronym: PROVERB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP211005
Record Dates: First submitted 2022-01-24; First posted 2022-09-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Revascularization
Keywords: Heart Failure; Multi-vessel disease; coronary artery bypass grafting; percutaeous coronary intervention
MeSH Terms: conditions — Heart Failure | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Open label, Blinded Endpoint, parallelgroup, active controlled, non-inferiority, multicenter trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor: The individual who evaluates the outcome(s) of interest
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angioplasty (Experimental): percutaneous coronary angioplasty with drug eluting stent implantation.
  Interventions: Procedure: Percutaneous coronary intervention
- Coronary artery bypass grafting (Active Comparator): Coronary artery bypass grafting has been chosen as the comparator because it is currently the reference strategy for revascularization in patients with multi-vessel disease and heart failure (ESC guidelines). Coronary artery bypass grafting technique will be total arterial revascularization unless internal mammary grafts are unavailable or have inadequate flow. All patients will be treated with anti-thrombotic therapy according to the European Society of Cardiology guidelines.
  Interventions: Procedure: Coronary artery bypass grafting

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — The studied intervention will be percutaneous coronary angioplasty with drug eluting stent implantation. Percutaneous coronary intervention may be performed during one single procedure or during staged procedures. The decision will be left at the investigator choice. PCI will be performed using drug eluting stent exclusively. The techniques for bifurcation lesions and chronic total occlusion angioplasty will be left at the operator choice. The choice of the drug eluting stent used will be left at the operator's choice. Anti-platelet therapy will be given to all patients randomized to PCI. The choice of the anti-thrombotic regiment and its duration will be left at the investigator choice (after assessment of initial presentation, bleeding and ischemic risks) but will have to comply with the European Society of Cardiology guidelines.
  Arms: Angioplasty
Procedure: Coronary artery bypass grafting — Coronary artery bypass grafting technique will be total arterial revascularization unless internal mammary grafts are unavailable or have inadequate flow. All patients will be treated with anti-thrombotic therapy according to the European Society of Cardiology guidelines
  Arms: Coronary artery bypass grafting

SUMMARY:
A short description, 5000 characters Ischemic cardiomyopathy related to coronary artery disease is currently the leading cause of heart failure. When it is responsible for heart failure, the coronary artery disease likely involves 2 or 3 vessels. Percutaneous coronary angioplasty, which is the other available technique for coronary revascularization, has never been evaluated in this indication. The results of retrospective registries studying the strategy for multivessel revascularization in patients with heart failure are inconsistent and no randomized study has been performed so far. Currently, ESC guidelines recommends to perform coronary-artery bypass grafting (IB) or percutaneous coronary intervention (IIa C) with the acknowledgement that percutaneous coronary intervention has never been properly evaluated in this setting. However, it has been previously demonstrated that left ventricle dysfunction significantly increases mortality and morbidity during and after cardiac surgery (3-10% mortality when LVEF is ≤30%). Moreover, the technical progresses in stent development and manufacturing have led to a dramatic decrease in the incidence of stent thrombosis and in-stent restenosis. Therefore, we hypothesize that percutaneous coronary angioplasty may be an attractive strategy for revascularization in patients with multi-vessel disease and left ventricle dysfunction, who are at high risk of surgical complication. Thus, we aim to test the hypothesis that percutaneous coronary intervention is non-inferior to coronary-artery bypass grafting for revascularization in patients with multivessel disease and left ventricle dysfunction.

The main objective is to demonstrate that percutaneous coronary angioplasty is non-inferior to coronary-artery bypass grafting for multivessel revascularization in patients with left ventricular dysfunction on major cardiac and cerebrovascular events (MACCE).

Method:A Prospective Randomized Open label, Blinded Endpoint, parallel-group, active controlled, non-inferiority, multicenter trial.

DETAILED DESCRIPTION:
Patients meeting the selection criteria will be enrolled after providing written informed consent. Patients will be randomized, in a 1:1 ratio, to receive either percutaneous coronary intervention with drug eluting stent or coronary-artery bypass grafting.

Whichever technique the patient is randomized to, revascularization will aim to be complete and both techniques will be performed following current guidelines and local practices. No myocardial viability assessment will be mandatory prior to inclusion. Both revascularization strategy will be associated with optimal medical therapy for heart failure.

Follow-up will be performed at 3, 12, 24, 36 and for patients enrolled in the trial early in the inclusion period, also at 48 months, and for all patients at the end of the study (3 years after inclusion of the last patient).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Left ventricle ejection fraction ≤35% measured by echocardiography, cardiac magnetic resonance imaging ventriculogram or gated Single Photon Emission Computed Tomography ventriculogram
* Multivessel disease suitable for revascularization:

  * Three vessel disease
  * Two vessel disease involving left main or proximal left anterior descending artery
* Clinical and anatomic eligibility for both percutaneous coronary intervention (PCI) and Coronary artery bypass grafting (CABG) as agreed to by the local Heart Team (interventionalist determines PCI appropriateness and eligibility; cardiac surgeon determines surgical appropriateness and eligibility)
* Ability to sign informed consent and comply with all study procedures, including follow-up for at least two years
* Affiliation to health insurance

Exclusion Criteria:

* Prior:

  * PCI of any coronary artery lesions within 6 months prior to randomization
  * CABG at any time prior to randomization
* Ongoing cardiogenic shock at the time of coronary angiogram (SBP< 90 mmHg with clinical signs of low output or patients requiring inotropic agents)
* Contra indication for PCI or CABG determined by the heart team
* Indication for another cardiac surgery (i.e. valvular surgery, aortic repair…) if CABG is performed
* ST elevation myocardial infarction < 30 days
* Non-cardiac illness with a life expectancy of less than 24 months
* Current participation in other investigational drug or device studies
* Women who are pregnant or nursing
* Females of childbearing potential without effective method of birth control
* Patients who are under tutorship or curatorship
* Patient on AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2030-07-16 (Estimated); Study Completion 2033-07-16 (Estimated)

PRIMARY OUTCOMES:
MACE | 3 years
  Comparison of MACE between PCI and CABG. Major adverse cardiac and cerebrovascular events (MACE) is a composite of death from any cause, stroke, myocardial infarction and unplanned hospitalization for heart failure or urgent revascularization.
MACE | 4 years
  Comparison of MACE between PCI and CABG.major adverse cardiac and cerebrovascular events (MACE) is a composite of death from any cause, stroke, myocardial infarction and unplanned hospitalization for heart failure or urgent revascularization.
MACE | 2 years
  Comparison of MACE between PCI and CABG. Major adverse cardiac and cerebrovascular events (MACE) is a composite of death from any cause, stroke, myocardial infarction and unplanned hospitalization for heart failure or urgent revascularization.
MACE | 1 year
  major adverse cardiac and cerebrovascular events (MACE) is a composite of death from any cause, stroke, myocardial infarction and unplanned hospitalization for heart failure or urgent revascularization.
MACE | 3 months
  Comparison of MACE between PCI and CABG
MACCE | an average of 54 months
  The composite outcome of death from any cause, stroke, myocardial infarction, unplanned hospitalization for heart failure or urgent revascularization or ischemia driven revascularization at the end of follow-up

SECONDARY OUTCOMES:
Death | an average of 54 months
  Death from any cause at the end of follow-up
Stroke | an average of 54 months
  Stroke at the end of follow-up
Myocardial Infarction | assessed up to 54 months
  Myocardial Infarction at the end of follow-up
Unplanned hospitalization | an average of 54 months
  Unplanned hospitalization at the end of follow-up
Ischemia driven revascularization | an average of 54 months
  Ischemia driven revascularization at the end of follow-up
Left ventricle ejection fraction | 1 year
  Left ventricle ejection fraction measure by echocardiography at 1 year
Heart Failure Questionnaire | 1 year
  Health Related Quality of life at 1 year
Treatment Burden Questionnaire | 1 year
  Treatment burden at 1 year (assessed using the Treatment Burden Questionnaire (TBQ))
Economic evaluation | an average of 54 months
  Economic evaluation incremental Cost-utility and cost effectiveness ratios

CONTACTS AND LOCATIONS:
Overall Officials: Akim SOUAG, Study Chair — Assistance Publique Hôpitaux de Paris- CHU Henri-Mondor; Romain GALLET, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris- CHU Henri-Mondor
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No